CLINICAL TRIAL: NCT00928486
Title: A Safety Confirmation Study On Lenalidomide With Dexamethasone In Japanese Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-022
Record Dates: First submitted 2009-06-09; First posted 2009-06-26 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and Dexamethasone (Experimental): Lenalidomide 25mg by mouth (PO) once daily (QD) on Days 1-21 of each 28 day cycle; When creatinine (CrCl) clearance <60 mL/min, the initial dose was 10mg and the dose could be increased to 15mg after 2 cycles if the investigator judged therapeutic effect was insufficient and tolerability was acceptable. Dexamethasone 40 mg by PO once QD on days 1-4, 9-12 and 17-20 of each 28 day cycle for the first 4 cycles and Days 1-4 for the remaining cycles beginning at Cycle 5.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 25mg PO for (days 1 - 21) of a 28-day cycle
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — Dexamethasone 40 mg by mouth (PO) daily (QD) on days 1-4, 9-12 and 17-20 of each 28 day cycle
  Other Names: Decadron

SUMMARY:
To evaluate the safety and efficacy of lenalidomide with dexamethasone in Japanese patients with previously treated multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign the informed consent form
* Age ≥ 20 years at the time of signing the informed consent form
* Subjects with previously treated multiple myeloma defined as follows:

  * Subjects must have received at least 1 prior anti-myeloma drug treatment regimen; and
  * Considered to have progression of disease (PD) that occurred either during or following the completion of the last anti-myeloma treatment regimen utilized prior to enrollment into this study
* Measurable levels of M-protein in serum (greater than or equal to 0.5 g/dL [5g/L]) or urine (greater than or equal to 0.2 g excreted in a 24-hour collection sample)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Must be able to adhere to the study visit schedule and other protocol requirements
* Females of childbearing potential (FCBP) must agree to use one or more of the following forms of contraception or abstain from heterosexual contact completely and have the male partners use a condom on the occasion of heterosexual contact in the following periods below:

  * For at least 28 days before starting study drug (in particular, the subject must abstain from heterosexual contact for 2 weeks prior to prescribing lenalidomide).
  * During the treatment phase (including the dose withholding period) For at least 28 days after the discontinuation/completion of the study drug (Methods of contraception)
  * Birth control pills
  * Intrauterine device (IUD)
  * Bilateral tubal ligation (FCBP must be referred to a health care provider who is familiar with contraceptive methods, if needed).
* Male subject must agree to use a condom during sexual contact with female irrespective of pregnancy potential
* Subjects must agree that study drug must be immediately discontinued, if pregnancy or a positive pregnancy test does occur in a female study subject or the partner of a male study subject during study participation

Exclusion Criteria:

* Pregnant or lactating females
* Subjects with a history of acute myocardial infarction within the past 6 months before starting the study drugs
* Subjects with any history or concurrent conditions of deep vein thrombosis or pulmonary embolus within the past 3 years before starting study drugs
* Subjects with tuberculous diseases, herpes simplex keratitis, systemic mycosis or other active infectious diseases
* Subjects with non-controlled diabetes, hypertension, digestive ulcer or glaucoma
* Subjects with posterior subcapsular cataracts
* Subjects with peripheral neuropathy of ≥Grade 2
* Subjects with any history or concurrent conditions which the Principal Investigator / subinvestigators consider inappropriate for participation in this study, and subjects with a serious disease or a mental disease, which is considered to become more risky if the subjects participate in this study.
* Subjects with a history of desquamative (blistering) rash while taking thalidomide
* Subjects with a history of using lenalidomide
* Subjects who have used thalidomide within 28 days before starting the study drugs
* Subjects with a history of hypersensitivity to dexamethasone
* Subjects who discontinued treatment due to grade 3 or 4 toxicity from high dose dexamethasone
* Subjects with a surgical wound after a visceral surgery performed recently
* Subjects who have undergone radiation therapy within 14 days before starting the study drugs
* Subjects who have used a chemotherapeutic agent, an immunomodulating agent or a study drug (a drug not commercially available) intended for the treatment of multiple myeloma (MM) within 28 days before starting the study drug
* Subjects with any history or concurrent conditions of malignancies, other than MM, unless the subject has been free of the disease for 3 years:

  * Basal cell carcinoma of the skin,
  * Squamous cell carcinoma of the skin,
  * Carcinoma in situ of the cervix,
  * Carcinoma in situ of the breast,
  * Incidental histologic finding of prostate cancer Tumor, Lymph Nodes, Metastasis (TNM) stage of T1a or T1b)
* Known human immunodeficiency virus (HIV) infection or HIV-1 positivity
* Subjects who have been diagnosed as an hepatitis b virus (HBV) carrier
* Subjects who are applicable to any of the following abnormal laboratory findings:

  * Absolute neutrophil count : < 1,000 /μL (1.0×10^9 /L)
  * Platelet count: <75,000 /μL (75×10^9 /L)
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT): > 3.0 times the upper limit of the standard range
  * Creatinine clearance: < 30 mL/min

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04-28 (Actual); Primary Completion 2010-09-10 (Actual); Study Completion 2010-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Takatoku, MD, Study Director — Celgene KK
Locations (8):
- Japan (8):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka Red Cross Hospital, Osaka, Osaka
  - Tokushima University, Tokushima, Tokushima
  - Keio University Hospital, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide and Dexamethasone
Started | 25
Efficacy Evaluable (EE) | 24 (EE population = given at least 1 dose of study drug, evaluated for efficacy and met eligibility)
Completed | 15 (Completed = those who continued responding to treatment; upon marketing approval, given lenalidomide)
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Disease Progression | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Population = includes all participants who received at least one dose of study drug
Arm/Group | Lenalidomide and Dexamethasone
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  Japan | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAE)
Description: A TEAE was defined as any AE that started on or after the first dose of study drug, and within End of Study (EOS) (28 days after the last dose of study drug received). A serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability; is a congenital anomaly/birth defect; or constitutes an important medical event. The intensity of AEs were graded 1 to 5 according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. For all other AEs not described in the CTCAE criteria, the intensity was assessed by the investigator as mild grade (Grade 1), moderate (grade 2), severe (grade 3), life-threatening (grade 4) or death (grade 5)
Time Frame: Day 1 of study drug through 28 days after the last dose of study drug; maximum treatment duration was 60.3 weeks
Population: Safety population included all 25 participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Dexamethasone
Number analyzed (Participants) | 25
participants
  Any Adverse Event (AE) | 25
  Drug-Related AE | 25
  Grade 3-4 Adverse Event | 22
  Drug-Related Grade 3-4 AE | 21
  Serious Adverse Event (SAE) | 12
  Drug-Related SAE | 9
  AE Leading to Study Drug Discontinuation | 4
  Related AE Leading to Len/Dex Discontinuation | 2
  AE leading to dose reduction or interruption | 17
  Related AE leading to dose reduction/interruption | 16

2. Secondary Outcome: Myeloma Response Rate
Description: Overall myeloma response rate was determined by the investigator using the Myeloma Response Determination Criteria adapted from Bladé criteria. A responder is any patient who showed at least a partial response. Overall myeloma response rate is defined as the percentage of participants who achieved a Complete Response (CR), plus a Remission Response (RR), plus a Partial Response (PR). A CR is the disappearance of monoclonal paraprotein and maintained for ≥ 6 weeks. RR is a 75-99% reduction in the level of the serum monoclonal paraprotein compared to baseline; 90-99% reduction in 24-hr urinary light chain excretion. PR is a 50-74% reduction in the level of monoclonal paraprotein compared to baseline; 50-89% reduction in 24-hr urinary light chain excretion.
Time Frame: From the time of the first dose of study drug to study completion; median duration on study was 42.1 weeks
Population: Efficacy Population = all participants who received at least one dose of study drug, who were evaluated for efficacy at least once after study drug dose administration and who met inclusion criteria
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Dexamethasone
Number analyzed (Participants) | 24
percentage of participants | 62.5

3. Secondary Outcome: Kaplan-Meier Estimates of Duration of Response (DoR)
Description: Duration of response was defined as the time from the first observation of a response (CR, RR or PR) to the first documented disease progression or relapse. For participants who did not progress during the study, duration of response was censored at the last adequate response assessment showing evidence of no disease progression. Disease progression is defined as an increase in M-protein serum monoclonal paraprotein and/or urine paraprotein or evidence of bone marrow plasmacytosis and plasma cells, an appearance of new or existing soft tissue plasmacytomas, an appearance of new or existing lytic bone lesions and/or hypercalcemia >11.5mg/dL
Time Frame: From the time of the first dose of study drug to study completion; the median duration on study was 42.1 weeks
Population: Efficacy Population = all participants who received at least one dose of study drug, who were evaluated for efficacy at least once after study drug dose administration and who met inclusion criteria who were responders
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide and Dexamethasone
Number analyzed (Participants) | 15
weeks | NA [NA to NA] — The median duration of response estimate was not reached at the last time data was censored at the last assessment date with no evidence of progression.

ADVERSE EVENTS:
Time Frame: Day 1 of study drug through 28 days after the last dose of study drug; maximum treatment duration was 60.3 weeks
Arm/Group | Lenalidomide and Dexamethasone
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (N=25)
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myocardial infarction (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Amyloidosis (Immune system disorders) | 1
Herpes zoster (Infections and infestations) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Diplegia 1 ( 4.0) (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (N=25)
Neutropenia (Blood and lymphatic system disorders) | 20
Lymphopenia (Blood and lymphatic system disorders) | 16
Leukopenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 7
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 4
Influenza (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Fibrin D dimer increased (Investigations) | 6
Blood glucose increased (Investigations) | 5
Fibrin degradation products increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
C-reactive protein increased (Investigations) | 2
Dysgeusia (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Hypogeusia (Nervous system disorders) | 2
Malaise (General disorders) | 7
Face oedema (General disorders) | 3
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 2
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Palpitations (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 2
Conjunctivitis (Eye disorders) | 2
Hot flush (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements varied; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.